CLINICAL TRIAL: NCT04230590
Title: Health Outcomes Via Positive Engagement in Schizophrenia (HOPE-S)
Brief Title: Health Outcomes Via Positive Engagement in Schizophrenia
Acronym: HOPE-S
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: MOH Office for Healthcare Transformation Pte. Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019/00720
Record Dates: First submitted 2019-12-30; First posted 2020-01-18 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia Spectrum Disorders
Keywords: Schizophrenia; Digital phenotyping; Relapse
MeSH Terms: conditions — Schizophrenia; Recurrence | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with schizophrenia spectrum disorders: Within 8 weeks post discharge from hospitalization at the Institute of Mental Health
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Participants will not receive any study intervention.
  During the 24-week study period, participants will complete five assessment visits and passive digital data from participant's smartphone and study-provided wrist wearable device will be collected.

SUMMARY:
This is an observational study where digital, clinical and health utilization data are collected from individuals with schizophrenia spectrum disorders who have been recently discharged from a psychiatric hospitalization. The data will be used towards building a model/algorithm capable of monitoring mental health and predicting adverse clinical events, such as relapse and re-admissions.

DETAILED DESCRIPTION:
In this research, participants will attend 6-weekly follow-up research visits (Weeks 0, 6, 12, 18, 24) over 24 weeks where clinical symptoms, cognition, functioning and well-being will be assessed. Passive digital data from smartphones and wrist wearable devices (e.g. sleep patterns, heart rate, location variance and entropy, phone usage frequency and duration, finger taps, ambient light, and physical activity) will be collected continuously during the 24 weeks. Audio recorded follow-up phone calls will be made to participants who consented to the optional audio recorded component at Weeks 3, 9, 15, 21. This study will also carry out an administrative follow-up at Week 24/termination and Week 52 to obtain healthcare utilization information (e.g. scheduled or unscheduled appointments, readmission, etc) since study enrollment.

Study findings will shed light on the relationship between digital biomarkers with clinical status and health utilization outcomes, as well as explore the feasibility and acceptability of digital sensors.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female aged 21 to 65 years (inclusive) at time of informed consent
* Has capacity to give informed consent
* Able to understand and comply with instructions in English
* Diagnosis of schizophrenia spectrum disorders assessed using the Structured Clinical Interview for DSM Disorders (SCID)
* Discharged patients from IMH (within 8 weeks post-discharge from IMH)

Exclusion Criteria:

* Female who is currently pregnant or planning a pregnancy within 6 months
* Has any other clinically significant medical condition or circumstance that, in the opinion of the Investigator, could affect participant safety, preclude evaluation of response, interfere with the ability to comply with study procedures, or prohibit completion of the study
* Has visual or physical motor impairment that could interfere with study tasks

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must be diagnosed with schizophrenia spectrum disorders and are within 8 weeks post discharge from hospitalization at the Institute of Mental Health.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression scale - Severity | up to 24 weeks
  A single item measuring severity of illness at the point of assessment relative to a clinician's experience with patients of the same diagnosis on a 7-point scale; a higher rating indicates greater severity.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | Week 0, 6, 12, 18, 24
  A 30-item clinical scale measuring positive symptoms, negative symptoms and general psychopathology. A higher total score indicates greater symptom severity.
Brief Negative Symptom Scale | Week 0, 24
  A 13-item scale that measures five negative symptom domains (blunted affect, alogia, asociality, anhedonia and avolition) and a subscale on Lack of Normal distress. Higher total score indicates greater negative symptoms.
Calgary Depression Scale for Schizophrenia | Week 0, 6, 12, 18, 24
  CDSS is a scale designed for the assessment of depression in schizophrenia, which differentiates between depression and the negative and positive symptoms of schizophrenia. Higher total score reflects greater severity.
Clinical Global Impression scale - Improvement | Week 6, 12, 18, 24
  A single item which measures how much the patient's illness has improved or worsened relative to a baseline state on a 7-point scale. A higher rating indicates greater worsening of illness.
Brief Adherence Rating Scale | Week 0, 6, 12, 18, 24
  A clinician-administered instrument to assess oral antipsychotic medication adherence of outpatients with schizophrenia. Greater proportion of doses taken in the past month indicate greater adherence (range: 0%-100%).
Columbia Suicide Severity Rating Scale | Week 0, 6, 12, 18, 24
  A scale assessing both suicidal ideation and behaviour.
Social and Occupational Functioning Assessment Scale | Week 0, 6, 12, 18, 24
  A scale designed to evaluate an individual's level of social and occupational functioning; its rating is not directly influenced by the overall severity of the individual's psychological symptoms. A greater rating reflects superior functioning in various areas of life (range: 0-100).
Brief Assessment of Cognition in Schizophrenia | Week 0, 24
  A cognitive battery which assesses attention, verbal and working memory, motor and processing speed, verbal fluency, reasoning and problem solving. Higher composite score indicates better cognitive function.
5-level EQ-5D | Week 0, 12, 24
  A standardized instrument developed as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. A higher score indicates best health imagined (range: 0-100).
Subjective Well-being under Neuroleptics scale - short form | Week 0, 24
  A self-rated instrument to assess well-being from a patient's perspective based on their subjective experiences during antipsychotic treatment. Higher total score indicates greater well-being.
Acceptability questionnaire | Week 24 or termination visit
  This questionnaire consists of an item measuring participants' satisfaction based on their experience of using digital devices on a scale range of 1 (Strongly disagree) to 7 (Strongly agree). Two other qualitative items in this questionnaire gather feedback on the strengths and suggested improvements for the system and user satisfaction.
Healthcare Utilization | 12 months
  Data from IMH's medical records which document events such as scheduled appointments, defaults, E-room attendances and hospitalizations will be used to explore healthcare utilization and its relationship with digital biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Lee, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore

REFERENCES:
- [Derived] Abdul Rashid NA, Martanto W, Yang Z, Wang X, Heaukulani C, Vouk N, Buddhika T, Wei Y, Verma S, Tang C, Morris RJT, Lee J. Evaluating the utility of digital phenotyping to predict health outcomes in schizophrenia: protocol for the HOPE-S observational study. BMJ Open. 2021 Oct 20;11(10):e046552. doi: 10.1136/bmjopen-2020-046552. PMID 34670760